CLINICAL TRIAL: NCT05642637
Title: Biobank Cycle Collection Study From Women Trying to Conceive
Brief Title: Biobank Cycle Collection
Acronym: BCC
Status: Active, not recruiting | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-1388
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy
Keywords: Fertility; Trying to Conceive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Early morning urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study will provide daily urine samples from volunteers who are trying to conceive in order to maintain the SPD biobank.

Study volunteers, seeking to conceive will be provided with a CE marked Clearblue Ovulation product to help them pinpoint their most fertile time and aid conception. All volunteers will provide daily early morning urine samples throughout the study period and keep a study diary of menses and pregnancy test results for up to 3 menstrual cycles.

Urine samples will be received in the clinical laboratory and aliquoted and stored at -80˚C until required.

DETAILED DESCRIPTION:
The purpose if this study is to maintain the SPD Biobank with urine samples from cycles in which conception occurred and ones where conception did not occur, together with associated sample information including demographic and clinical data e.g. menses days, volunteer age and reproductive hormone concentrations.

Study volunteers, seeking to conceive will be recruited to the study after providing written informed consent. All volunteers will be provided with a CE marked Clearblue Ovulation product to help them pinpoint their most fertile time and aid conception and be required to collect daily early morning urine samples throughout the study until pregnancy is confirmed or their next menstrual period starts. Volunteers will be required to keep a daily diary of menses, sample collection and pregnancy test results. The study will last for up to 3 consecutive menstrual cycles.

Urine samples will be received in the clinical laboratory and will be tested for the presence of hormones related to pregnancy and fertility, then aliquoted and stored in the SPD Biobank at -80˚C until required for product development or evaluation purposes.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 and over actively trying to conceive
* At least 2 regular consecutive cycles since last pregnancy/miscarriage/ stopping breastfeeding or contraception
* Willing to disclose their pregnancy status and provide urine samples.
* Willing to give informed consent and comply with the study procedures

Exclusion Criteria:

* Trying to conceive for >6 months (under 35 years) or > 3 months (35 years and over)
* Has a diagnosis of Polycystic Ovary Syndrome (PCOS)
* Taking medication or has known condition which means they should not get pregnant.
* Currently pregnant or breastfeeding
* Using any treatment which may affect the menstrual cycle (e.g. contraceptive pill)
* Using or has previously used infertility medications or hormone replacement medications containing LH or hCG \ (e.g. Pregnyl®)
* Using or undergoing any other medical treatment for fertility such as ovulation drugs, artificial insemination and assisted fertility such as IVF or ICSI
* Peri-or post-menopausal, e.g. experiencing symptoms: irregular menstrual periods, hot flushes, night sweats, sleep disturbances and/or moods swings
* Abnormal liver or kidney function
* Taking antibiotics containing tetracycline.
* Participated in this study within the last 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women trying to conceive
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Collection of daily urine samples from women trying to conceive | 3 years
  Daily samples collected throughout the cycle in which conception occurs

CONTACTS AND LOCATIONS:
Overall Officials: Raniero Zazzeroni, Study Director — SPD Development Company
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No